CLINICAL TRIAL: NCT06217861
Title: An Open-Label, Dose-Escalation and Dose-Expansion Phase I Clinical Study to Evaluate the Tolerability, Safety and Efficacy of VGM-R02b in Patients With Glutaric Acidemia Type I
Brief Title: A Study to Evaluate the Tolerability, Safety and Efficacy of VGM-R02b
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Vitalgen BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGM-R02b-101; 2023LP01348 (Other: CDE)
Record Dates: First submitted 2023-12-12; First posted 2024-01-23 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-01

CONDITIONS: Glutaric Acidemia Type I; Glutaric Aciduria Type I
Keywords: AAV; gene therapy; ICV; GCDH
MeSH Terms: conditions — Glutaric Acidemia I

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VGM-R02b (Experimental): VGM-R02b is an adeno-associated viral vector 9 delivering human Glutaryl-CoA Dehydrogenase (GCDH) gene.
  Interventions: Biological: VGM-R02b

INTERVENTIONS:
Biological: VGM-R02b — Administered as specified in the treatment arm.
  Other Names: rAAV9-GCDH

SUMMARY:
Phase I, open-label, single-arm, single-dose, trial of VGM-R02b (gene replacement therapy) in patients with Glutaric Acidemia Type I (GA-I) who meet enrollment criteria and are genetically confirmed by GCDH gene mutation. 1 to 3 patients aged≤ 6 years at the time of screening will be enrolled in each dose group in the dose escalation part. In the dose expansion part, the sample size will be statistically calculated and adjusted according to the efficacy and safety data in the dose escalation part.

DETAILED DESCRIPTION:
This study consists of screening period, treatment period and postoperative monitoring period and follow-up period. During the screening period (Days -28 to -1), patients whose parent(s)/legal guardian(s) provide informed consent will complete screening procedures to determine eligibility for trial enrollment. Eligible subjects will be admitted to the clinical research center before surgical administration to complete the preoperative examination and determine the surgical plan. Ommaya fluid reservoir capsule implantation will be used in this study (if there were problems with Ommaya implantation, intra-cerebroventricular injection could also be used for drug administration). The day of administration set to be D1. Prophylactic immunosuppressive therapy including Methylprednisolone, Prednisolone and Rapamycin was initiated on D1. Then all the examinations during the 7-day postoperative observation period will be completed based on the evaluation time point specified in the Schedule of Assessments table. Subjects may be discharged 7 days after the infusion, based on Investigator judgment. During the outpatient follow-up period (up to 52 weeks after administration), subjects will return at regularly scheduled intervals for efficacy and safety assessments until the End of Trial. After the End of Trial visit, eligible patients will be asked to participate into the long-term follow up trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be ≤ 6 years;
2. History of diagnosis of GA-I, and confirmed by gene mutation analysis with biallelic GCDH mutation;
3. At the time of screening, there was one of the obvious neurological manifestations associated with the following diseases, including macrocephaly, dystonia, and motor/intellectual development Poor fertility, epilepsy, abnormal EEG;
4. Those who are receiving standard treatment recommended by the guidelines and whose symptoms remain poorly controlled by the investigator;
5. Plasma GA and 3-OHGA levels were higher than the normal range during screening;

Exclusion Criteria:

1. Participation in gene therapy or stem cell transduction therapy at any time prior to screening for this trial or participation in any other clinical trial within 3 months prior to screening;
2. Recurrent seizures that are not suitable for surgery, based on Investigator judgment;
3. Current severe liver or kidney or cardiovascular disease or coagulation dysfunction, autoimmune deficiency, or uncontrolled autoimmune disease or need immunosuppressive long-term treatment, poorly controlled diabetes (HBA1C ≥7% at screening) or high blood pressure;
4. Active viral infection (includes HIV or serology positive for hepatitis B or C or syphilis);
5. Presence or history of malignancy;
6. Received systemic immunosuppressive therapy within 3 months prior to screening;
7. Received vaccine within 4 weeks prior to administration or plan to receive vaccine within 1 year after administration;
8. Plan to receive surgery during the study;
9. Current using medications including, drugs, herbal or OTC medications that strongly inhibit or induce CYP3A4 or P-glycoprotein (P-gp), e.g., metoclopramide, grapefruit juice, ketoconazole, erythromycin;
10. Abnormal brain structure, not suitable for lateral ventricle administration;
11. Abnormal laboratory test results, which are judged by the investigator not suitable for surgery;
12. History of systemic hypersensitivity reaction to investigational product, the excipients contained in the formulation, or prophylactic immunosuppressant;
13. Contraindicated use of corticosteroids and sirolimus;
14. Contraindicated with general anesthesia or sedation;
15. As judged by the investigator, unable to perform lateral ventricle puncture or Ommaya capsule implantation or lumbar puncture;
16. Unable to perform CT or MRI;
17. Poor compliance;
18. Any other situation where, judged by the investigator, the subject is not suitable for participating in this study.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of AEs and SAEs | up to 52 weeks
  An AE is any untoward medical occurrence (eg any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
Evaluate changes from baseline in vital signs, and clinical laboratory results | up to 52 weeks
  Clinically significant abnormal laboratory values or test results must be identified through a review of values outside of normal ranges/clinically notable ranges, significant changes from baseline or the previous visit, or values which are considered to be non-typical in participant with the underlying disease.

SECONDARY OUTCOMES:
Changes in Barry Albright Dystonia Scale from baseline. | up to 52 weeks
  The BAD Scale is a 5-point, criterion-based, ordinal scale designed to assess dystonia in eight body regions: eyes, mouth, neck, trunk, and the four extremities. Raters score dystonia as none (0), slight (1), mild (2), moderate (3), or severe (4).
Changes in Peabody Developmental Motor Scale (PDMS-2) from baseline. | up to 52 weeks
  The Peabody Developmental Motor Scales, a norm referenced tool commonly used to assess infants' fine and gross motor development, also is widely used for children of preschool age.
Changes in Bayley Scales of Infant and Toddler Development (BSID) or Wechsler Preschool and Primary Scale of Intelligence (WPPSI) from baseline. | up to 52 weeks
  BSID is an extensive formal developmental assessment tool for diagnosing developmental delays in early childhood, this will be used in 1~42 month patients.
  The WPPSI uses subtests to determine a child's Verbal and Performance IQ scores as well as the processing speed for children ages over 42 months.
Neuroimaging. | up to 52 weeks
  Changes in clinically significant abnormalities on brain MRI and MRS compared to Baseline.
Biomarkers. | up to 52 weeks
  Changes of C5DC GA, 3-OHGA in CSF and plasma.
Immunogenicity. | up to 52 weeks
  The antibody titer and the number of subjects with positive anti-AAV9 and anti-hGCDH antibodiesin the blood and CSF.
  The antibody titer and the number of subjects with positive anti-AAV9 and anti-hGCDH specific T cell immune response of peripheral blood mononuclear cells (PBMC).

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Shu, Principal Investigator — The Children's Hospital Zhejiang University Shcool of Medicine; Rulai Yang, Principal Investigator — The Children's Hospital Zhejiang University Shcool of Medicine; Guanping Dong, Principal Investigator — The Children's Hospital Zhejiang University Shcool of Medicine
Locations (1):
- The Children's Hospital Zhejiang University Shcool of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers when VGO-Cm01 is fully approved.